CLINICAL TRIAL: NCT00003553
Title: A Phase II Study of HLA-Matched Peripheral Blood Mobilized Hematopoietic Progenitor Cell Transplantation for Metastatic Renal Cell Carcinoma Followed by Allogeneic T-Cell Infusion as Adoptive Immunotherapy
Brief Title: Peripheral Stem Cell Transplant in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Richard W. Childs, National Heart, Lung, and Blood Institute
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 970196; NHLBI-97-H-0196; CDR0000066610 (Other: NIH); NCT00001635 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: patients with progressive metastatic renal cell carcinoma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): The target for progenitor cell is >=5 x 106 CD 34/kg.
  Interventions: Other: HLA Matched Peripheral BLood Stem Cells

INTERVENTIONS:
Other: HLA Matched Peripheral BLood Stem Cells — Cell Product

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as cyclophosphamide and fludarabine, before a donor peripheral blood stem cell transplant helps stop the growth of tumor cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining tumor cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine with or without mycophenolate mofetil or methotrexate after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well peripheral stem cell transplant works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effect of allogeneic peripheral blood stem cell transplantation (PBSCT) in patients with metastatic renal cell carcinoma.
* Evaluate the safety and toxicity of a nonmyeloablative, low-intensity, preparative regimen followed by an HLA-matched allogeneic PBSCT in these patients.
* Determine engraftment by measuring donor-recipient chimerism in lymphoid and myeloid lineages in patients treated with this regimen.
* Determine the relationship between donor-host chimerism and the incidence of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the effect of lymphocyte infusions on donor-host chimerism in this patient population.
* Determine the response rate, disease-free survival, overall survival, and mortality from the procedure or tumor progression in patients treated with this regimen.

OUTLINE:

* Nonmyeloablative preparative regimen: Patients receive 1 of 3 preparative regimens prior to peripheral blood progenitor cell (PBPC) transplantation. (Regimens 2 and 3 closed to accrual as of 10/1/03.)

  * Regimen 1: Patients receive cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine IV over 30 minutes on days -5 to -1.
  * Regimen 2 (closed to accrual as of 10/1/03): Patients receive cyclophosphamide IV over 1 hour on days -7 and -6, fludarabine IV over 30 minutes on days -5 to -1, and antithymocyte globulin on days -5 to -2.
  * Regimen 3 (closed to accrual as of 10/1/03): Patients receive cyclophosphamide IV over 1 hour on days -8 to -6, fludarabine IV over 30 minutes on days -5 to -1, and antithymocyte globulin on days -5 to -2.
* PBPC transplantation: Patients undergo mobilized CD34+ PBPC transplantation on day 0. PBPC transplantation may be repeated on days 1 and 2, if deemed necessary.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive 1 of 3 GVHD prophylaxis regimens.

  * Regimen 1 (closed to accrual as of 10/17/00): Patients receive cyclosporine IV over 12 hours or orally beginning on day -4 and continuing for up to approximately 3 months.
  * Regimen 2 (open to accrual from 10/17/00 through 2/11/02): Patients receive cyclosporine as in regimen 1. Patients also receive mycophenolate mofetil.
  * Regimen 3 (open to accrual as of 2/11/02): Patients receive cyclosporine as in regimen 1. Patients also receive methotrexate.
* Donor lymphocyte infusions: Patients with progressive disease on days 15-30, day 60, or day 100, without GVHD, receive infusion(s) of donor lymphocytes. Further donor lymphocyte infusions after day 100 may be given at the discretion of the attending physician.

Patients are followed every 2 months for 6 months, every 3 months for 2 years, and then every 6 months for 2½ years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA - PATIENT:

Ages 18-80 years.

Biopsy proven metastatic RCC, not amenable to complete surgical resection, progressive bidimensionally evaluable clinically or radiographically.

No prior treatment for RCC within 30 days.

HIV negative.

ECOG performance status of 1 or less.

No major organ dysfunction precluding transplantation.

DLCO greater than or equal to 65% predicted.

Left ventricular ejection fraction greater than or equal to 40%.

HLA 6/6 or 5/6 matched family related donor available.

Ability to comprehend the investigational nature of the study and provide informed consent.

Durable power of attorney signed.

INCLUSION CRITERIA - DONOR:

HLA 6/6 or 5/6 matched family related donor.

Fit to receive G-CSF and give peripheral blood stem cells (normal blood counts, normotensive, no history of stroke).

Ability to comprehend the investigational nature of the study and provide informed consent.

Ages 18-80.

EXCLUSION CRITERIA (any of the following) - PATIENT:

Patient Pregnant.

Age greater than 80 or less than 18 years.

ECOG performance status of 2 or more. Psychiatric disorder or mental deficiency of the patient or donor sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

Major anticipated illness or organ failure incompatible with survival from BMT where survival is considered insufficient to assess transplant outcome (i.e. less than 3 months).

DLCO less than 65% predicted.

Left ventricular ejection fraction less than 40%.

Serum creatinine greater than 2.5mg/dl or creatinine clearance less than 50 cc/min by 24 hour urine collection.

Serum bilirubin greater than 4 mg/dl, transaminases greater than 3 x upper limit of normal.

HIV positive.

History of other malignancies except basal cell or squamous carcinoma of the skin.

Disease which is limited and amenable to complete surgical resection.

Lack of evidence for progressive disease.

Disease which is not evaluable clinically or radiographically.

Evidence for CNS metastatic disease.

Disease involving greater than 25% of the liver radiographically.

Hypercalcemia (greater than 2.5 mmol/L).

EXCLUSION CRITERIA - DONOR:

Donor pregnant or lactating.

Donor HIV or HBsAg positive.

History of malignancy within 5 years except basal cell or squamous carcinoma of the skin.

Donor unfit to receive G-CSF and undergo apheresis (Uncontrolled hypertension, history of stroke, thrombocytopenia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 1998-02-09 (Actual); Primary Completion 2011-06-27 (Actual); Study Completion 2011-06-27 (Actual)

PRIMARY OUTCOMES:
The anti-tumor effect of allogenic peripheral blood stem cell transplantation in patients with progressive metastatic renal cell carcinoma. | 5 Years

SECONDARY OUTCOMES:
Evaluate the safety and toxicity of a nonmyeloblative, low intensity, preparative regimen followed by an HLA matched allogenic peripheral blood stem cell transplant in patients with metastatic renal cell carcinoma. | 100 Days
The relationship between donor-host chimerism and the incidence of acute and chronic GVHD. The effect of donor lymphocyte infusions on donor-host chimerism. Response rate, disease free and overall survival and mortality. | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Childs, MD, Study Chair — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- NIH - Warren Grant Magnuson Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Carvallo C, Geller N, Kurlander R, Srinivasan R, Mena O, Igarashi T, Griffith LM, Linehan WM, Childs RW. Prior chemotherapy and allograft CD34+ dose impact donor engraftment following nonmyeloablative allogeneic stem cell transplantation in patients with solid tumors. Blood. 2004 Feb 15;103(4):1560-3. doi: 10.1182/blood-2003-04-1170. Epub 2003 Oct 9. PMID 14551148
- [Result] Childs R, Chernoff A, Contentin N, Bahceci E, Schrump D, Leitman S, Read EJ, Tisdale J, Dunbar C, Linehan WM, Young NS, Barrett AJ. Regression of metastatic renal-cell carcinoma after nonmyeloablative allogeneic peripheral-blood stem-cell transplantation. N Engl J Med. 2000 Sep 14;343(11):750-8. doi: 10.1056/NEJM200009143431101. PMID 10984562